CLINICAL TRIAL: NCT05816577
Title: Safety and Viability of an E. Coli Nissle Colibactin Knockout in Healthy Volunteers
Acronym: SECONI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Max Nieuwdorp (Other)
Responsible Party: Sponsor-Investigator, Max Nieuwdorp, Prof. dr., Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL83158.018.22
Record Dates: First submitted 2023-03-09; First posted 2023-04-18 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Diabetes
Keywords: advanced microbiome therapeutics; diabetes; safety
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, controlled, safety study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomised through Castor (eCRF). Treatment allocation is blinded for investigators and participants. The pharmacist has access to the randomisation list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EcN (Active Comparator): E Coli Nissle wildtype 10^11 once daily for 7 days
  Interventions: Dietary Supplement: E Coli Nissle
- EcN colibactin-knockout (Experimental): EcN colibactin-knockout 10^11 once daily for 7 days
  Interventions: Dietary Supplement: EcN Colibactin knockout

INTERVENTIONS:
Dietary Supplement: EcN Colibactin knockout — E coli Nissle strain with ClbP-gene removed and therefore not producing colibactin
  Arms: EcN colibactin-knockout
Dietary Supplement: E Coli Nissle — E Coli wildtype strain
  Arms: EcN

SUMMARY:
E. coli Nissle (EcN) is a well-established human probiotic. However, it has been found that it produces colibactin, linked to colorectal cancer. In this safety trial, the safety and properties of a novel, colibactin-knockout EcN strain (EcNΔClbP) is investigated.

DETAILED DESCRIPTION:
In this randomised controlled intervention study, the investigators will compare EcN vs. EcN colibactin-knockout (EcNΔClbP), given once daily for 7 days, in a population of healthy individuals. Safety will be established using adverse event reporting, study visits and laboratory parameters. Pharmacokinetics will be established at the beginning and the end of the study. EcN/EcNΔClbP gut engraftment properties and effects on gut microbiome composition will be assessed using fecal analyses (qPCR, shotgun metagonmics). In addition, effects on glucose homeostasis will be studied using continuous glucose monitoring.

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female of Caucasian descent

  * If female, postmenopausal
* Age: 18-65 years old
* BMI: 18-25 kg/m2
* Subjects should be able to give informed consent

Exclusion Criteria:

* Use of any systemic medication (except for paracetamol), including proton pump inhibitors, antibiotics and pro-/prebiotics in the past three months or during the study period.
* Use of the EcN probiotic strain (Mutaflor®) in the past 12 months.
* (Expected) prolonged comprised immunity (e.g. due to recent cytotoxic chemotherapy or human immunodeficiency viruses (HIV) infection with a CD4-T cell count < 240/mm3).
* History of moderate to severe disease of the digestive tract, such as celiac disease, chronic diarrhoea (≥3 stools/day for >4 weeks), chronic obstipation (<2 defecations/week for >3 months), Irritable Bowel Syndrome (IBS) (according to Rome IV criteria) or Inflammatory Bowel Disease (IBD).
* Any gastro-intestinal disorder within the past 6 months
* Smoking or illicit drug use (e.g. amphetamine/cocaine/heroin/GHB) in the past three months or use during the study period.
* Use of >21 units of alcohol per week on average in the past three months or use of >2 units of alcohol during the study period.
* Simultaneous participation in other studies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Adverse events | 3 weeks
  The number, duration and severity of adverse reactions to assess the safety/tolerability of the EcNΔClbP strain compared to the wild type strain.
CRP | Weekly, during 3 weeks
  Changes in CRP (mg/L)
Leucocytes | Weekly, during 3 weeks
  Changes in leucocytes (10^9/L)
Renal function | Weekly, during 3 weeks
  Changes in renal function, expressed as kreatinin levels (micromol/L) throughout the study
Bilirubin | Weekly, during 3 weeks
  Changes in bilirubin in micromol/L throughout the study
alkaline phosphatase | Weekly, during 3 weeks
  Changes in alkaline phosphatase in U/L throughout the study
gamma-GT in U/L | Weekly, during 3 weeks
  Changes in gamma-GT in U/L throughout the study
AST | Weekly, during 3 weeks
  Changes in AST in U/L throughout the study
ALT | Weekly, during 3 weeks
  Changes in ALT in U/L throughout the study
Hemoglobin | Weekly, during 3 weeks
  Changes in hemoglobin in mmol/L throughout the study
trombocytes | Weekly, during 3 weeks
  Changes in trombocytes in 10^9/L throughout the study
eosinophils | Weekly, during 3 weeks
  Changes in eosinophils in 10^9/L throughout the study
basophils | Weekly, during 3 weeks
  Changes in basophils in 10^9/L throughout the study
neutrophils | Weekly, during 3 weeks
  Changes in neutrophils in 10^9/L throughout the study
monocytes | Weekly, during 3 weeks
  Changes in monocytes in 10^9/L throughout the study
Lipid profile | Weekly, during 3 weeks
  Changes in lipid profile throughout the study
Homeostatic model of insulin resistance (HOMA-IR) | Weekly, during 3 weeks
  Changes in HOMA-IR throughout the study
Gastro-intestinal quality of life - questionnaire | Weekly, during 3 weeks
  Changes in Gastro-intestinal quality of life (GIQLI) score. The maximum score is 155, the minimum score is 31. A higher score represents a better outcome.
Bristol Stool Chart | Weekly, during 3 weeks
  Changes in Bristol Stool Chart score throughout the study. Stools can be scored from 1 (hard stool) to 7 (watery stool). A score of 4 is considered ideal.

SECONDARY OUTCOMES:
Number of copies of EcN (qPCR) | Daily during 2 weeks
  Quantification of EcN in faeces samples collected throughout the two weeks via quantitative polymerase chain reaction (qPCR)
Microbiome composition | Weekly during 3 weeks
  Comparison of relative abundances of species throughout the study using shotgun metagenomics

OTHER OUTCOMES:
Fecal 24h bile acids | Weekly during 3 weeks
  Changes in 24h faecal bile acids will be measured at V2, V3 and V4.
Fasting blood bile acids | Weekly during 3 weeks
  Changes in fasting plasma bile acids will be measured at V2, V3 and V4.
Fecal 24h short chain fatty acids | Weekly during 3 weeks
  Changes in 24h faecal and fasting and short-chain fatty acids will be measured at V2, V3 and V4.
Fasting blood short chain fatty acids | Weekly during 3 weeks
  Changes in fasting short-chain fatty acids will be measured at V2, V3 and V4.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No